CLINICAL TRIAL: NCT06295003
Title: Impact of COVID-19 Pandemic on Headache Evaluations in the Pediatric Emergency Department
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Alberto Cappellari, Principal investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: CEFA-COVID
Record Dates: First submitted 2024-03-04; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; Headache Disorders; Emergency Service, Hospital
MeSH Terms: conditions — COVID-19; Headache Disorders; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Background: To evaluate the impact of COVID-19 on evaluations in the pediatric emergency department (ED) because of headache as main symptom.

Methods: Number and clinical features of patients evaluated in the pediatric ED of a single site in Milan,Italy, were collected between January 2017 and January 2022. The impact of COVID-19 on evaluation rates was quantified by using the incidence rate ratio (IRR) and 95% confidence intervals (CI) between the pandemic (March 2020 to January 2022) and the prepandemic period (January 2017 to February 2020).

ELIGIBILITY:
Inclusion Criteria:

* range of age: 2 - 18 years
* sex: all
* headache as main symptom

Exclusion Criteria:

* headache in the context of head trauma, because of different diagnostic-care in Pediatric Emergency Department

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: patients aged 2-18 years evaluated in Pediatric Emergency Department because of headache as main symptom
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
During the study period, 890 evaluations were registered: the number of partecipants was 689 over the prepandemic period and 201 over the pandemic period. Mean age at evaluation was 10 years (range: 1 to 17 years). | the pandemic (March 2020 to January 2022) and the prepandemic period (January 2017 to February 2020).

SECONDARY OUTCOMES:
Evaluation rates per month were 18.1 during the prepandemic period and 8.7 during COVID-19 pandemic, with peaks in autumn and winter and drops in summer. The reduction in evaluation rate was higher for secondary headache when compared with primary one | the pandemic (March 2020 to January 2022) and the prepandemic period (January 2017 to February 2020).

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Emergency Department Clinica de Marchi, Foundation IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy